CLINICAL TRIAL: NCT03311074
Title: Methodology Study to Investigate the Utility of Retroviral Insertion Site Analysis in Samples From Subjects Treated With Strimvelis™ Gene Therapy
Brief Title: Retroviral Insertion Site Methodology Study
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Replaced with new observational study design
Sponsor: Fondazione Telethon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STRIM-002
Record Dates: First submitted 2017-10-11; First posted 2017-10-16 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2023-11

CONDITIONS: Immune System Diseases
Keywords: Sonication Linker Medicated Polymerase Chain Reaction; Previously GSK2696273; Gene therapy; Adenosine deaminase deficiency; Retroviral insertion site; Severe combined immunodeficiency; Strimvelis
MeSH Terms: conditions — Immune System Diseases; Severe combined immunodeficiency due to adenosine deaminase deficiency; Severe Combined Immunodeficiency

STUDY DESIGN:
Intervention Model Description: There will be no separate treatment groups in the study.
Masking Description: No masking will be performed in the study and all subjects who have received Strimvelis, either in previous clinical trials or as a registered product, will be included in the analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Strimvelis treatment receivers (Experimental): Approximately 15 subjects with ADA-SCID who were previously received Strimvelis will be included in the analysis and a total of 5 blood samples will be collected from each subject at approximately annual interval.
  Interventions: Genetic: Strimvelis

INTERVENTIONS:
Genetic: Strimvelis — Strimvelis is a gene therapy that aims to restore ADA function in hematopoietic cell lineages and prevent the immunological manifestations. Strimvelis is a cluster of differentiation (CD) 34+ cell enriched dispersion of human bone marrow derived hematopoietic stem cells for infusion which have been transduced with a retroviral vector containing the human ADA gene.

SUMMARY:
Adenosine deaminase (ADA) is an enzyme involved in the development and functioning of the immune system. Deficiency of ADA results in severe combined immunodeficiency (SCID), a fatal inherited immune disorder. Strimvelis is a gene therapy that aims to insert ADA function into blood cells and halt or reverse the conditions caused by decreased ADA enzyme levels, such as impaired immune function. It is important to consider long term follow-up of patients who have received Strimvelis, including evaluation of the risk of insertion near certain genes that may lead to unexpected activation of those genes (oncogenesis). The objective of this study is to evaluate the use of a new technique to identify where Strimvelis has become inserted in the genetic sequence, and potential implications for patient care. This new technique is known as sonication linker mediated polymerase chain reaction (SLiM-PCR) for retroviral insertion site (RIS) analysis. The study will recruit at least 15 pediatric or adult patients with ADA-SCID who have been treated with Strimvelis, either in previous clinical trials or as a registered product. Recruitment for the study may remain open for up to 2 years even if 15 subjects are recruited sooner. Study participation will last for up to 5 years. A total of 5 blood samples will be collected from each subject at approximately annual intervals.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, pediatric or adult, subjects with ADA-SCID, who have been previously treated with Strimvelis.
* Capable of giving signed informed consent or signed informed consent provided by the subject's parent or legal guardian.

Exclusion Criteria:

* Presence of concomitant condition(s) that in the Investigator's opinion makes participation in the study unsuitable or may prevent compliance with the protocol requirements.
* Unlikely to comply with the requirements of the protocol (i.e. attendance for blood sampling on an approximately annual basis).
* Transportation of viable samples to the European Union (EU) central laboratory from the subject's home country is not possible.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06-25 (Actual); Primary Completion 2020-07-09 (Actual); Study Completion 2020-07-09 (Actual)

PRIMARY OUTCOMES:
Mean abundance measurement | Up to 5 years
  The accuracy and precision of SLiM-PCR methodology will be assessed using whole blood samples, taken from subjects treated with Strimvelis, spiked with control insertion site deoxyribonucleic acid (DNA). The mean abundance will be calculated between subjects at every time point, within subjects over time points and between the same sample within a time point within a subject.
Coefficient of variation measurement | Up to 5 years
  The accuracy and precision of SLiM-PCR methodology will be assessed using whole blood samples, taken from subjects treated with Strimvelis, spiked with control insertion site DNA. The coefficient of variation will be calculated between subjects at every time point, within subjects over time points and between the same sample within a time point within a subject.

SECONDARY OUTCOMES:
Measurement of clone abundance of more than 5 percent | Up to 5 years
  Abundance of clones in subject's samples will be measured by SLiM-PCR, where abundance estimates will be derived from the number of individual sheared DNA fragments and the number of DNA barcodes in the linker sequences.
Shannon diversity index measurement | Up to 5 years
  The Shannon diversity index is an index that is commonly used to characterize species diversity in a community. The diversity of the clones in subject's samples will be determined using Shannon diversity. Shannon diversity index will be summarized using mean and coefficient of variation.

CONTACTS AND LOCATIONS:
Overall Officials: Fondazione Telethon, Study Director — Fondazione Telethon